CLINICAL TRIAL: NCT05171959
Title: Characterization of the Platelet and Immune Response in Adults Receiving SARS-CoV-2 Vaccine
Brief Title: Platelet and Immune Response in Covid-19 Vaccine
Acronym: Vax-SPEED-IT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Lucia Stefanini (Unknown); Stefania Basili (Unknown)
Responsible Party: Principal Investigator, Roberto Cangemi, Prof. Roberto Cangemi, University of Roma La Sapienza
Other Study IDs: PLTCOVAX
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV-2 Vaccination
Keywords: SARS-CoV-2; Covid-19; Vaccine; Platelets; Immunity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anticoagulated whole blood, serum, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 mRNA vaccines, administered with a two-dose regimen, have been shown to provide protection against Covid-19. However, the thromboinflammatory response toward these vaccines has never been explored as they exploit a completely new technology. It was reported that mRNA vaccines are highly reactogenic right after vaccine administration in particular in young adults, but we do not know which cells drive the early immune response to LNP-mRNA vaccines in humans and if platelets become activated as well. Moreover, it is not known if female, who have a heightened immune response to other vaccines, are able to mount a faster response to this new type of vaccines.

Objectives of the study is to characterize the platelet and immune response and the platelet-immune cross-talk in subjects undergoing SARS-CoV-2 vaccination.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a systemic, potentially severe and life-threatening disease, triggered by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Since the first cases of SARSCoV-2 infection were officially diagnosed, in December 2019, more than 280 million cases and 5 million deaths have been declared worldwide. In response to this public health emergency the international scientific community has made an enormous effort to understand the virus and to develop a safe vaccine to prevent the spread of COVID-19. Just few days after the World Health Organization declared the SarsCoV-2 outbreak a global pandemic, it was published the structure of the Spike viral protein [1], which has provided critical clues to design vaccines. Within less than 12 months several vaccines against SARS-CoV-2 have been developed. The first vaccine that has been approved in Europe and that is already being administered in Italy is the COVID-19 RNA vaccine, developed by BioNTech-Pfizer (BNT162b2). Both this vaccine and the one developed by Moderna consist of a lipid nanoparticle (LNP) that deliver a nucleoside-modified messenger RNA (mRNA) encoding the precise genetic information of the immunogen (SARS-CoV-2 full-length spike protein) to antigen presenting cells and elicits potent immune responses. mRNA is transiently expressed, does not integrate into the genome, and is degraded by physiological pathways.mRNA vaccines are molecularly well defined, synthesized efficiently from DNA templates by in vitro transcription, which is cell- and animal-origin material-free. mRNA production and LNP formulation are fast processes of high scalability, rendering this technology suitable for rapid vaccine development and pandemic vaccine supply [2].

Both mRNA vaccines, administered with a two-dose regimen, have been shown to provide a 94-95% protection against Covid-19 in persons 16 years of age or older [3,4]. However, the thromboinflammatory response toward these vaccines has never been explored as they exploit a completely new technology. For instance, it was reported that mRNA vaccines are highly reactogenic right after vaccine administration in particular in young adults [3], but we do not know which cells drive the early immune response to LNP-mRNA vaccines in humans and if platelets become activated as well. Moreover, it is not known if female, who have a heightened immune response to other vaccines, are able to mount a faster response to this new type of vaccines.

AIMS OF THE STUDY

Primary objective To characterize the platelet and immune response and the platelet-immune cross-talk in subjects undergoing SARS-CoV-2 vaccination.

Secondary objective To study the short-term kinetics of the immune and the antibody response in subjects undergoing SARS-CoV-2 vaccination.

STUDY PROTOCOL

We will enrol female and male (1:1) volunteers without signs of infection who will be subjected to SARS-CoV-2 Vaccination.

Enrolled healthy volunteers will be asked to undergo venous blood withdrawals at the following time-points:

* T0: 0-24 hours before the first dose of the vaccine;
* T1: 72±24 hours after the first dose of vaccine administration;
* T2: 10±2 days after first dose of vaccine administration;
* T3: 0-24 hours before the second dose of vaccine;
* T4: 72±24 hours after second dose of vaccine administration;
* T5: 10±2 days after second dose of vaccine administration.

A small aliquot of blood anticoagulated with sodium citrate will be used within 1 hour from blood withdrawal to perform in vivo assays (see list below), the rest will be centrifuged within 2 hours and plasma and serum samples will be stored at -80°C for further analysis (see list below).

REFERENCES

1. Wrapp D, Wang N, Corbett KS, Goldsmith JA, Hsieh CL, Abiona O, Graham BS,McLellan JS.Cryo-EM structure of the 2019-nCoV spike in the prefusion conformation. Science. 2020 Mar 13;367(6483):1260-1263. doi:10.1126/science.abb2507.
2. Pardi N, Hogan MJ, Porter FW, Weissman D. mRNA vaccines - a new era in vaccinology. Nat Rev Drug Discov. 2018 Apr;17(4):261-279. doi:10.1038/nrd.2017.243.
3. Polack FP, Thomas SJ, Kitchin N, et al. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020;383(27):2603-2615. doi:10.1056/NEJMoa2034577
4. Anderson EJ, Rouphael NG, Widge AT, Jackson LA, et al.; mRNA-1273 Study Group. Safety and Immunogenicity of SARS-CoV-2 mRNA-1273 Vaccine in Older Adults. N Engl J Med. 2020 Dec 17;383(25):2427-2438. doi: 10.1056/NEJMoa2028436.
5. Lanza GA, Barone L, Scalone G, et al.; Inflammation-related effects of adjuvant influenza A vaccination on platelet activation and cardiac autonomic function. J Intern Med. 2011 Jan;269(1):118-25. doi: 10.1111/j.1365-2796.2010.02285.x.

At baseline (T0) each adult enrolled will be asked to fill in a short questionnaire, to provide information on baseline characteristics, previous relevant medical history (i.e. chronic medical conditions, use of drugs with a particular focus on immunosuppressant agents), smoking and exposure to SARS-CoV-2 (i.e. if a previous diagnosis of COVID-19 was received).

At any further timepoint (T1-T4), each participant will be asked to fill in a short questionnaire on symptoms related to vaccination, occurrence of COVID-19 infection, and drugs used, to account for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers without signs of SARS-CoV2 infection who will be subjected to SARS-CoV-2 Vaccination

Exclusion Criteria:

* Anti-platelet or anti-coagulant medications in the past 10 days
* Autoimmune disease
* Reported severe immunosuppression
* Pregnancy or breastfeeding
* Recent transfusions of platelets or plasma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enrol 32 female and male (1:1) volunteers without signs of infection who will be subjected to SARS-CoV-2 Vaccination.
  Enrolled healthy volunteers will be asked to undergo venous blood withdrawals at the following time-points:
  * T0: 0-24 hours before the first dose of the vaccine;
  * T1: 72±24 hours after the first dose of vaccine administration;
  * T2: 10±2 days after first dose of vaccine administration;
  * T3: 0-24 hours before the second dose of vaccine;
  * T4: 72±24 hours after second dose of vaccine administration;
  * T5: 10±2 days after second dose of vaccine administration.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Platelet-leukocytes aggregates quantification | 6 months
  Percentage of platelet-leukocytes aggregates (PLA) among blood leukocytes. PLA are identified based on the expression of CD41a in the individual leukocyte subpopulations.

SECONDARY OUTCOMES:
Cytokine Array in plasma | 6 months
  Plasmatic inflammatory cytokine concentrations (including IL-1β, IFN-α2, IFN-γ, TNF-α, IL-6, IL-8, IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33 and MCP-1) will be analysed using commercial bead-based immunoassay.
Detection of Circulating SARS-Cov-2 Neutralization Antibodies | 6 months
  Serum SARS-CoV-2 neutralizing antibodies will be detected using COVID-19 Immunorank™ MICRO-ELISA (Leinco Technologies, Inc St. Louis MO).
Platelet Phenotypic and Functional Analysis | 6 months
  Expression of surface receptors and platelet activation in whole anticoagulated blood (in vivo assays)
Soluble markers of platelet activation: sP-selectin, sCD40L. | 6 months
  Plasma sP-selectin and sCD40 analysed will be analysed by commercial ELISA kits.
Pro-Inflammatory Chemokines | 6 months
  CCL8, MCP-1, CXCL10, CCL11, CCl17, CCL5, CCL3, CXCL9, CXCL5, CCL20, CXCL5, CCL20, CXCL1, CXCL11, CCL4 will be analysed with commercial kits.
Immunophenotyping | 6 months
  % of neutrophils, eosinophils, classical/nonclassical monocytes, CD4+T cells, CD8+Tcell, B cells, Treg cells, NK cells, NKT cells in whole anticoagulated blood.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cangemi, MD, Principal Investigator — University of Roma La Sapienza; Stefania Basili, MD, Study Chair — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided